CLINICAL TRIAL: NCT01090154
Title: Certolizumab Pegol for the Treatment of Moderate to Severe Ulcerative Colitis: An Open Label Study
Brief Title: Study of Cimzia for the Treatment of Ulcerative Colitis
Acronym: UC CIMZIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: UCB Pharma (Industry); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Scott Lee, Associate Professor, Medicine/Division of Gastroenterology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37823; CZP-UC-001 (Other: Protocol Number)
Record Dates: First submitted 2010-03-15; First posted 2010-03-19 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; UC; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cimzia (Experimental): Treatment with open label Cimzia (certolizumab pegol)
  Interventions: Drug: Cimzia

INTERVENTIONS:
Drug: Cimzia — Cimzia 400mg administered via two 200mg subcutaneous injections at weeks 0, 2, and 4; followed by every 4 week dosing.
  Other Names: certolizumab pegol

SUMMARY:
The purpose of this study is to determine if Cimzia (certolizumab pegol) is an effective treatment for patients with Ulcerative colitis.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease which often results in significant morbidity as well as impairment in quality of life. Cimzia (certolizumab pegol), an inhibitor of tumor necrosis factor-alpha, is an effective treatment for Crohn's disease, a similar inflammatory bowel disease. The aims of this study are to determine if Cimzia is effective for both the induction and maintenance of response/remission for the patients with moderate to severe Ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria

1. Adults aged 18-75 years
2. Established diagnosis of UC (by routine clinical, radiologic, endoscopic, and histologic criteria) of at least 3 months duration
3. Moderate to severe active disease, defined by Mayo score > 6 with endoscopic subscore > 2
4. Ability to understand the study protocol and treatments, willingness to comply with all study requirements, and ability to provide informed consent
5. No history of prior tuberculosis (TB), no signs or symptoms of active TB, and negative Quantiferon gold test or PPD and chest X-ray showing no active or latent TB at screening or within the 6 months prior to the screening visit.
6. Screening blood tests must meet the following criteria: white blood cell count > 3000/µL (with neutrophils > 1500/µL and lymphocytes > 500/µL), hemoglobin > 8 g/dL, platelet count > 100,000/µL, liver function tests < 3 times the upper limit of normal, serum creatitine < 1.5 mg/dL
7. Screening stool sample negative for Clostriduim difficile, ova & parasites, and aerobic pathogens, including Aeromonas, Plesiomonas, Salmonella, Shigella, Yersinia, Campylobacter, and E. coli spp.
8. Medication use must meet the following criteria:

   1. Rectally administered topical 5-aminosalicylates (5-ASAs)/corticosteroids: must be discontinued by 1 month prior to baseline; not allowed during the study
   2. Oral 5-ASAs: allowed if at stable dose for at least 2 weeks prior to baseline; can remain on this stable dose during the study
   3. Antibiotics for UC: must be discontinued by 1 month prior to baseline; not allowed during the study
   4. Antidiarrheals: must be discontinued by 2 weeks prior to baseline; not allowed during the study
   5. Corticosteroids: allowed if at Prednisone dose equivalent of 20 mg/d or less, stable for 2 weeks prior to baseline (dose/taper during study discussed below); budesonide is allowed at a dose less than or equal to 9 mg/day if at stable dose for 2 weeks prior to baseline
   6. 6-Mercaptopurine (6MP)/Azathioprine/Methotrexate: allowed if on for at least 8 weeks, at stable dose for at least 4 weeks prior to baseline; can remain on this stable dose during the study
   7. Anti-TNF therapy: Patients must be naive to CZP. Patients may have had prior exposure to anti-TNF therapy (e.g., infliximab, adalimumab, golimumab), however patients who are primary non-responders to more than one anti-TNF medication are excluded. Patients must have been off their prior anti-TNF medication for at least 8 weeks prior to baseline.
   8. Integrin inhibitor therapy: Patients may have had prior exposure to integrin inhibitor therapy (e.g., vedolizumab). Patients must have been off of integrin inhibitor therapy for at least 8 weeks prior to baseline.
   9. Cyclosporine: patients previously receiving Cyclosporine for UC must have been off their prior Cyclosporine therapy for at least 4 weeks prior to baseline.
   10. Any other medications for the treatment of Ulcerative colitis or investigational medications: must be discontinued at least 1 month or 5 half-lives (whichever is longer) before baseline; not allowed during the study
9. Female subjects of childbearing potential must agree to practice an effective method of birth control during the study and for 12 weeks after the last dose of study drug. Acceptable methods include: oral contraceptives, transdermal contraceptives, injectable contraceptives, implants, intrauterine devices, barrier methods with spermicide, or surgical sterility.

Exclusion Criteria

1. Diagnosis of Crohn's disease or indeterminate colitis, or clinical findings suggestive of Crohn's disease
2. Fulminant disease, toxic megacolon, or anticipated imminent colectomy
3. Presence of ileal pouch or ostomy
4. Pregnancy, desire to become pregnant during the following 18 months, or breast feeding
5. Surgery of any kind within 2 months of screening or anticipated surgery of any kind during the study
6. Anticipated imminent hospitalization for any medical conditions
7. Active ongoing infection of any kind
8. Current use of total parenteral nutrition
9. History of:

   1. Congestive heart failure or significant coronary artery disease (including myocardial infarction, percutaneous coronary intervention, or coronary artery bypass within 6 months of screening)
   2. Cancer
   3. Colonic dysplasia (except sporadic adenomas). Also, patients found to have colonic dysplasia at any time during the study will be withdrawn from the study.
   4. HIV, chronic or active hepatitis B or C, or patients considered at high risk for these infections (obtained by history/detailed medical chart review except for hepatitis B, which will be tested for with blood sample)
   5. Prior opportunistic infection within 6 months of screening or prior opportunistic infection while on other anti-TNF therapy
   6. Hepatic disease (cirrhosis, chronic active hepatitis, or LFT abnormalities as above)
   7. Renal insufficiency (see above)
   8. Clinically important pulmonary disease (as determined subjectively)
   9. Demyelinating disease
   10. Organ transplantation, including bone marrow (except corneal)
   11. Lymphoproliferative disorder

SAMPLE SIZE CALCULATION

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of patients achieving clinical response determined by patient reported symptoms and investigator's assessment of mucosal healing via endoscopy measured by Total Mayo Score at Week 14 compared to Week 0. | Week 14
  Clinical response is defined as a decrease in the Total Mayo Score of at least 3 points by Week 14 compared to Week 0.

SECONDARY OUTCOMES:
To determine the proportion of patients achieving clinical remission determined by patient reported symptoms and investigator's assessment of mucosal healing via endoscopy measured by Total Mayo Score at Week 14 compared to Week 0. | Week 14
  Clinical remission is defined as a total Mayo score of less than or equal to 2 with no individual subscore greater than 1 at Week 14 compared to Week 0.
To determine the proportion of patients achieving clinical response or clinical remission at week 54 per the same criteria as listed above. | Week 54
To determine the proportion of patients achieving mucosal healing at weeks 14 and 54 defined as a Mayo endoscopic subscore less than 2. | Week 14/54
To determine the corticosteroid-sparing effects of certolizumab pegol over a years treatment time. | Week 54
  To determine if patients are able to remain off steroids and maintain response or remission with certolizumab pegol alone and not necessitate concomitant treatment with steroids.
To determine the colectomy rate between week 0 and week 54 | Week 54
To determine the change in mean or median total or partial Mayo score between week 0 and week 54 | Week 54
To determine the change in mean or median serum CRP levels between week 0 and week 54 | Week 54
To determine the change in mean or median IBDQ or SIBDQ scores between week 0 and week 54 | Week 54
To determine all adverse events, serious adverse events, opportunistic infections, and injection site reactions between week 0 and week 64 | Week 64

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Lee, MD, Principal Investigator — University of Washington; Mark T Osterman, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No